CLINICAL TRIAL: NCT05210075
Title: Mindful With Your Baby for Mothers of Infants With (Parental) Stress in a Non-clinical Setting: A Wait-list Controlled Pilot Trial
Brief Title: Mindful With Your Baby in a Non-clinical Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Amsterdam (Other)
Responsible Party: Principal Investigator, Irena Veringa-Skiba MSc, MSc., University of Amsterdam
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015-CDE-4632
Record Dates: First submitted 2021-12-16; First posted 2022-01-27 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Stress Reduction

STUDY DESIGN:
Intervention Model Description: A wait-list controlled pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A wait list controlled (Experimental): A wait list controlled
  Interventions: Behavioral: Mindful with your Baby program

INTERVENTIONS:
Behavioral: Mindful with your Baby program — The training Mindful with your baby consists of eight weekly 2-h sessions, plus a follow-up session 8 weeks later. The first and the fifth sessions are with the mothers only. The rest of the sessions are with both mothers and babies present. The sessions are finished by explaining the new home practices. Home practice consists of reading handouts about mindfulness and mindful parenting for mothers with a baby, formal and informal meditation practice.

SUMMARY:
In this pilot waitlist-controlled trial, 17 mothers with infants (2-15 months) admitted themselves for a Mindful with your Baby (MwyB) training in a non-clinical setting because of (parental) stress. MwyB was offered in groups of three to six dyads and consisted of eight 2-hour sessions. Participants completed questionnaires on symptoms of parental stress, stress, depression, anxiety, mindfulness and self-compassion at 8-week waitlist, pretest, posttest and 8-week follow-up.

DETAILED DESCRIPTION:
This study used a quasi-experimental design. Participants were recruited in various ways. After admitting themselves to the study, participants were called by the trainer, to check inclusion criteria: a subjective experience of (parental) stress, and the ability to speak and read Dutch. Exclusion criteria were: a current unsafe situation for the baby, and maternal psychosis or suicidality. None of the mothers that admitted themselves were excluded. Participants gave informed consent online, before completing the first set of online questionnaires using forced responses via Qualtrics software. A waitlist assessment was administered 8 weeks prior to the start of the training, to control for the effects of time, assessment and other intervention. The pretest assessment took place in the week before the start of the training, posttest the week after the end of the training and follow-up eight weeks after the end of the training, respectively.

Intervention The MwyB training consists of 8 weekly 2-hour sessions, and a follow-up session 8 weeks after the last session. It is adapted to the presence of the babies (in 7 of the 9 sessions), and the themes that play a role for most mothers with a baby. The MwyB training was given and studied before from May 20213 until september 2016 in a clinical setting, given by a mental health psychologist/mindfulness/mindful parenting trainer plus an infant mental health specialist (study published in 2017, see citations). In this study the training was given in a non-clinical setting by a licensed midwife/mindfulness/mindful parenting/mindfulness based childbirth and parenting trainer plus an assistant (a master student Psychology or Pedagogics). The main role of the assistant was to ensure both physical and emotional safety of the babies during the meditation in which mothers closed their eyes. Four groups of 3 to 6 dyads were given between March 2016 and December 2017.

Measures

* Parental stress. Parental stress was assessed with the short form of the Dutch Parenting Stress Index, based on the American Parenting Stress Index.
* Symptoms of stress, depression, and anxiety. Maternal symptoms of stress, depression, and anxiety were assessed by a short form of the Depression Anxiety Stress Scales (DASS-21).
* Mindfulness. Mindfulness was assessed using the short form of the Dutch version of the five-facet mindfulness questionnaire. See citation.
* Self-compassion. To measure self-compassion the 3-item Self-Compassion Scale (SCS-3) was used.
* Acceptability. Acceptability was assessed by an evaluation questionnaire at posttest. An adapted version of the stress reduction program evaluation, developed at the Center for Mindfulness of the University of Massachusetts Medical School, was used. Session attendance rate, reported in the evaluation questionnaire, was calculated by dividing the number of attended sessions by the total number of sessions.

Data analyses

All outcomes were tested with multilevel regression models that are known to accommodate missing data and dependence between observations.

ELIGIBILITY:
Inclusion Criteria:

* a subjective experience of (parental) stress, and the ability to speak and read Dutch.

Exclusion Criteria:

a current unsafe situation for the baby, and maternal psychosis or suicidality.

Max Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Parental stress change from waitlist to start of intervention | The change between waitlist assessment at 8 weeks pre-intervention and 1 week pre-intervention assessment
  Short form of the Dutch Parenting Stress Index, minimum 1 (better), maximum 6 (worse)
Parental stress change from start of intervention until end of intervention | The change between 1 week pre-intervention assessment and 1 week post-intervention assessment.
  Short form of the Dutch Parenting Stress Index, minimum 1 (better), maximum 6 (worse)
Parental stress change from start of intervention until follow-up session | The change between 1 week pre-intervention assessment and 8 weeks post-intervention assessment.
  Short form of the Dutch Parenting Stress Index minimum 1 (better), maximum 6 (worse)
Change in symptoms of stress, depression, and anxiety from waitlist to start of intervention | The change between waitlist assessment at 8 weeks pre-intervention and 1 week pre-intervention assessment
  The Depression Anxiety Stress Scales, short form, minimum 0 (better), maximum 3 (worse)
Change in symptoms of stress, depression, and anxiety from start of intervention until end of intervention | The change between 1 week pre-intervention assessment and 1 week post-intervention assessment.
  The Depression Anxiety Stress Scales, short form, minimum 0 (better), maximum 3 (worse)
Change in symptoms of stress, depression, and anxiety from start of intervention until follow-up session | The change between 1 week pre-intervention assessment and 8 weeks post-intervention assessment.
  The Depression Anxiety Stress Scales, short form, minimum 0 (better), maximum 3 (worse)
Mindfulness change from waitlist to start of intervention | The change between waitlist assessment at 8 weeks pre-intervention and 1 week pre-intervention assessment
  The Dutch version of the five-facet mindfulness questionnaire, short form, minimum 1 (worse), maximum 5 (better) .
Mindfulness change from start of intervention until end of intervention | The change between 1 week pre-intervention assessment and 1 week post-intervention assessment.
  The Dutch version of the five-facet mindfulness questionnaire, short form, minimum 1 (worse), maximum 5 (better) .
Mindfulness change from start of intervention until follow-up session | The change between 1 week pre-intervention assessment and 8 weeks post-intervention assessment.
  The Dutch version of the five-facet mindfulness questionnaire, short form, minimum 1 (worse), maximum 5 (better) .
Self-compassion change from waitlist to start of intervention. | The change between waitlist assessment at 8 weeks pre-intervention and 1 week pre-intervention assessment
  3-item Self-Compassion Scale, minimum 1 (worse), maximum 7 (better)
Self-compassion change from start of intervention until end of intervention | The change between 1 week pre-intervention assessment and 1 week post-intervention assessment.
  3-item Self-Compassion Scale, minimum 1 (worse), maximum 7 (better)
Self-compassion change from start of intervention until follow-up session | The change between 1 week pre-intervention assessment and 8 weeks post-intervention assessment.
  3-item Self-Compassion Scale, minimum 1 (worse), maximum 7 (better)

IPD SHARING:
Plan to Share IPD: No
Data can be shared if a reasonable scientific request will be provided.

REFERENCES:
- [Background] Potharst ES, Aktar E, Rexwinkel M, Rigterink M, Bogels SM. Mindful with Your Baby: Feasibility, Acceptability, and Effects of a Mindful Parenting Group Training for Mothers and Their Babies in a Mental Health Context. Mindfulness (N Y). 2017;8(5):1236-1250. doi: 10.1007/s12671-017-0699-9. Epub 2017 Apr 13. PMID 28989548
- [Background] Loyd BH, Abidin RR. Revision of the Parenting Stress Index. J Pediatr Psychol. 1985 Jun;10(2):169-77. doi: 10.1093/jpepsy/10.2.169. No abstract available. PMID 4020601
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] de Bruin EI, Topper M, Muskens JG, Bogels SM, Kamphuis JH. Psychometric properties of the Five Facets Mindfulness Questionnaire (FFMQ) in a meditating and a non-meditating sample. Assessment. 2012 Jun;19(2):187-97. doi: 10.1177/1073191112446654. PMID 22589426
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717